CLINICAL TRIAL: NCT04686786
Title: A 57-Week, Multicenter, Active-treatment, Open-label Extension Trial of CVL-865 as Adjunctive Therapy in Adults With Drug-Resistant Focal Onset Seizures
Brief Title: An Open-label Extension Trial of CVL-865 as Adjunctive Therapy in the Treatment of Focal Onset Seizures
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed early after CVL-865-SZ-001 (NCT04244175) did not meet its primary objective
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-865-SZ-002; 2019-004057-83 (EudraCT Number)
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Seizures
Keywords: CVL-865; Anti-epileptic drugs (AEDs); PF-06372865; γ-aminobutyric acid (GABA); focal epilepsy; partial seizure
MeSH Terms: conditions — Seizures; Epilepsies, Partial | interventions — PF-06372865

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CVL-865 25 mg (Experimental): Participants will receive CVL-865 tablets orally twice daily (BID) up to the maximum dose of 25 milligrams (mg) until Week 57 during the treatment period.
  Interventions: Drug: CVL-865

INTERVENTIONS:
Drug: CVL-865 — Participants will receive 25 mg CVL-865 tablets orally BID during the treatment period. The dose may be decreased to 17.5 mg BID for tolerability.
  Other Names: PF-06372865

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of CVL-865 as adjunctive therapy in participants with focal onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed treatment in Trial CVL-865-SZ-001 (NCT04244175)
* A female participant of childbearing potential who is sexually active with a nonsterilized male partner must agree to use a highly effective method of contraception from signing of informed consent through 30 days post last dose
* A male participant with a pregnant or a nonpregnant partner of childbearing potential must agree to use a condom during treatment and until the end of relevant systemic exposure in the male participant for 94 days following the last dose with the investigational medicinal product (IMP)
* Participants who are capable of giving signed informed consent
* Participants who are able, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures

Exclusion Criteria:

* Participants who, in the opinion of the investigator, medical monitor, or sponsor, should not participate in the trial
* Participants who, in the judgment of the investigator, experienced poor tolerability to the IMP during the double-blind trial or whose safety assessments resulted in new concerns that would suggest that the participant may not be appropriate for 57 weeks of treatment with CVL-865 in an extension trial
* Participants who experienced status epilepticus during Trial CVL-865-SZ-001
* Participants who have demonstrated substantial noncompliance to trial procedures in Trial CVL-865-SZ-001, based on the investigator's judgment, would not be eligible for this trial
* Participants who answer "yes" on the C-SSRS Suicidal Ideation Item 4 or Item 5 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan, or Active Suicidal Ideation with Specific Plan and Intent), or participants who answer "yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior), or participants who, in the opinion of the investigator, present a serious risk of suicide
* Participants with any of the following abnormalities in clinical laboratory tests at Visit 1, as assessed by the central laboratory and confirmed by a single repeat measurement, if deemed necessary (Females: Hemoglobin <11 gram per deciliter (g/dL); Males: hemoglobin <12 g/dL; White blood cell (WBC) count <3.0 x 10 power 9 per liter (10^9/L); Neutrophil count <2.0 x 10^9/L; Platelet count <150 × 10^9/L)
* Participants who would be likely to require the use of prohibited concomitant medications during the trial
* Female participants who have a positive pregnancy test result

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (54):
- United States (25):
  - Little Rock, Arkansas, Little Rock, Arkansas
  - New Haven, Connecticut, New Haven, Connecticut
  - Gulf Breeze, Florida, Gulf Breeze, Florida
  - Jacksonville, Florida, Jacksonville, Florida
  - Miami Lakes, Florida, Miami Lakes, Florida
  - Orlando, Florida, Orlando, Florida
  - Port Charlotte, Florida, Port Charlotte, Florida
  - Tampa, Florida, Tampa, Florida
  - Honolulu, Hawaii, Honolulu, Hawaii
  - Lexington, Kentucky, Lexington, Kentucky
  - Scarborough, Maine, Scarborough, Maine
  - Baltimore, Maryland, Baltimore, Maryland
  - Bethesda, Maryland, Bethesda, Maryland
  - Boston, Massachusetts, Boston, Massachusetts
  - Chesterfield, Missouri, Chesterfield, Missouri
  - Saint Louis, Missouri, St Louis, Missouri
  - Hackensack, New Jersey, Hackensack, New Jersey
  - New York, New York, New York
  - Rochester, New York, Rochester, New York
  - Toledo, Ohio, Toledo, Ohio
  - Oklahoma City, Oklahoma, Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania, Philadelphia, Pennsylvania
  - Charleston, South Carolina, Charleston, South Carolina
  - Nashville, Tennessee, Nashville, Tennessee
  - Salt Lake City, Utah, Salt Lake City, Utah
- Australia (8):
  - Camperdown, New South Wales, Camperdown, New South Wales
  - Randwick, New South Wales, Randwick, New South Wales
  - Westmead, New South Wales, Westmead, New South Wales
  - Herston, Queensland, Herston, Queensland
  - Fitzroy, Victoria, Fitzroy, Victoria
  - Heidelberg, Victoria, Heidelberg, Victoria
  - Melbourne, Victoria, Melbourne, Victoria
  - Parkville, Victoria, Parkville, Victoria
- Poland (7):
  - Bydgoszcz, Kujawsko-Pomorskie, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Kraków, Malopolskie, Krakow, Lesser Poland Voivodeship
  - Gdańsk, Pomorskie, Gdansk, Pomeranian Voivodeship
  - Wojnicz, Lskie, Wojnicz, Wojnicz Lskie
  - Białystok, Bialystok
  - Warszawa, Warsaw
  - Lodz, Lodz, Łódź Voivodeship
- Serbia (2):
  - Kragujevac, Sumadija, Kragujevac, Sumadija
  - Neurology Department, Kragujevac, Kragujevac, Sumadija
- South Korea (2):
  - Gwangjin-gu, Seoul, Gwangju, Seoul
  - Irwon-Ro Gangnam-gu., Seoul, Irwon-dong, Seoul
- Spain (7):
  - Malaga,, Málaga, Andalusia
  - Barcelona, Catalunya, Barcelona, Catalonia
  - Barcelona, Catalonia, Barcelona, Catalonia
  - Terrassa, Catalonia, Terrassa, Catalonia
  - Madrid, Madrid
  - Sevilla, Seville
  - Valencia, Valencia
- Ukraine (3):
  - Uzhgorod, Uzhhorod, Uzhgorod
  - Kyiv, Kyiv
  - Lviv, Lviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurrell R, Iredale P, Evrard A, Duveau V, Ruggiero C, Roucard C. Pronounced antiseizure activity of the subtype-selective GABAA positive allosteric modulator darigabat in a mouse model of drug-resistant focal epilepsy. CNS Neurosci Ther. 2022 Nov;28(11):1875-1882. doi: 10.1111/cns.13927. Epub 2022 Aug 14. PMID 35965432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment into the trial consisted of eligible participants who completed the Maintenance Phase of Trial CVL-865-SZ-001 (NCT04244175).
Groups:
- CVL-865 25 mg: Participants received 25 milligrams (mg) CVL-865 tablets orally twice daily (BID).
Period: Overall Study
Arm/Group | CVL-865 25 mg
Started | 105
Received at Least 1 Dose of Investigational Medicinal Product (IMP) | 105
Completed | 39
Not Completed | 66
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Lack of Efficacy | 25
Not completed — Treatment with Prohibited Concomitant Medications | 1
Not completed — Study Terminated by Sponsor | 14
Not completed — Withdrawal by Subject | 15
Not completed — Other than specified | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received at least 1 dose of investigational medicinal product (IMP).
Groups:
- CVL-865 25 mg: Participants received 25 mg CVL-865 tablets orally BID.
Arm/Group | CVL-865 25 mg
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 87
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 3
  White | 90
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: A TEAE was defined as an AE that started after the first dose of IMP in the open-label trial or a previously reported AE that increased in intensity, became serious, trial drug-related, or resulted in death, discontinuation, interruption, of reduction of IMP after the first dose of IMP in the open-label trial. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in the 'Reported Adverse Events module'.
Time Frame: From first dose of study drug up to Week 61
Population: The Safety Set included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | CVL-865 25 mg
Number analyzed (Participants) | 105
Participants
  Participants with TEAE | 88
  Participants with TESAE | 11

2. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Electrocardiogram (ECGs)
Description: 12-lead ECGs recordings were obtained after the participant had been supine and at rest for at least 5 minutes. The number of participants with significant abnormalities is reported by 'change from baseline in QT interval as corrected for heart rate by Fridericia's formula (QTcF)'.
Time Frame: Baseline up to Week 57
Population: The Safety Set included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | CVL-865 25 mg
Number analyzed (Participants) | 105
Participants | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Measurements
Description: Vital signs were measured with the participant in a sitting/semi-recumbent position after 5 minutes rest and included temperature, systolic and diastolic blood pressure, and heart rate.
Time Frame: Baseline up to Week 57
Population: The Safety Set included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | CVL-865 25 mg
Number analyzed (Participants) | 105
Participants | 2

4. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Physical and Neurological Examination Results
Description: A complete physical examination consisted of measurement of weight and a review of the following body systems: head, ears, eyes, nose, mouth, skin, heart, lungs, lymph nodes, and gastrointestinal, genitourinary, and musculoskeletal systems. A full neurological examination included an assessment of the participant's mental status (level of consciousness, orientation, speech, memory, etc), cranial nerves, motor (muscle appearance, tone, strength, and reflexes), sensation (including Romberg sign), coordination, and gait. Reported here is the number of participants with clinically significant changes in physical or neurological examination results.
Time Frame: Baseline up to Week 57
Population: The Safety Set included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | CVL-865 25 mg
Number analyzed (Participants) | 105
Participants
  Number of participants with any clinically significant physical examination findings | 5
  Number of participants with any clinically significant neurological examination findings | 7

5. Primary Outcome: Suicidality Based on the Columbia Suicide-Severity Rating Scale (C-SSRS)
Description: The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).
Time Frame: Baseline up to Week 61
Population: The Safety Set included all participants who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | CVL-865 25 mg
Number analyzed (Participants) | 105
Participants
  Suicidal Ideation: (1) Wish to be dead | 6
  Suicidal Ideation: (2) Non-specific active suicidal thoughts | 5
  Suicidal Ideation: (3) Active suicidal ideation with any methods (not plan) without intent to act | 1
  Suicidal Ideation: (4) Active suicidal ideation with some intent to act, without specific plan | 2
  Suicidal Ideation: (5) Active suicidal ideation with specific plan and intent | 0

6. Primary Outcome: Change From End of Treatment in Modified Clinical Institute Withdrawal Assessment - Benzodiazepines (mCIWA-B) Score at the End of Post-treatment Follow-up (Week 61)
Description: The modified Clinical Institute Withdrawal Assessment - Benzodiazepines (mCIWA-B) is a sensitive instrument to measure withdrawal under conditions where there is a taper of medication (rather than abrupt discontinuation). It consists of 17-items that monitor the type and severity of benzodiazepine withdrawal symptoms such as irritability, fatigue, appetite, and sleeplessness. The total score ranges from 1 (no withdrawal) to 68 (extreme withdrawal) with higher scores indicating more severe withdrawal.
Time Frame: Week 57, Week 61
Population: The Safety Set included all participants who received at least 1 dose of IMP. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CVL-865 25 mg
Number analyzed (Participants) | 83
score on a scale | -1.4 (8.45)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the start of safety data collection to the end of the study. The median time on follow-up was 260 days.
Description: The Safety Set included all participants who received at least 1 dose of IMP.
Arm/Group | CVL-865 25 mg
All-Cause Mortality (participants affected / at risk) | 1/105
Serious Adverse Events (participants affected / at risk) | 11/105
Other Adverse Events (participants affected / at risk) | 77/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVL-865 25 mg (N=105)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
DIVERTICULITIS INTESTINAL PERFORATED (Infections and infestations) | 1 (1)
CRANIOFACIAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 2 (2)
STATUS EPILEPTICUS (Nervous system disorders) | 1 (1)
APATHY (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVL-865 25 mg (N=105)
NEUTROPENIA (Blood and lymphatic system disorders) | 11 (15)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 9 (22)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4)
CONSTIPATION (Gastrointestinal disorders) | 3 (4)
DIARRHOEA (Gastrointestinal disorders) | 5 (5)
NAUSEA (Gastrointestinal disorders) | 5 (7)
VOMITING (Gastrointestinal disorders) | 5 (5)
FATIGUE (General disorders) | 15 (16)
FEELING HOT (General disorders) | 3 (3)
NON-CARDIAC CHEST PAIN (General disorders) | 3 (5)
COVID-19 (Infections and infestations) | 8 (8)
EAR INFECTION (Infections and infestations) | 3 (3)
INFLUENZA (Infections and infestations) | 3 (3)
CONTUSION (Injury, poisoning and procedural complications) | 3 (5)
FALL (Injury, poisoning and procedural complications) | 13 (16)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 3 (3)
HEAD INJURY (Injury, poisoning and procedural complications) | 3 (4)
SKIN LACERATION (Injury, poisoning and procedural complications) | 3 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 4 (4)
WEIGHT DECREASED (Investigations) | 4 (4)
WEIGHT INCREASED (Investigations) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5)
ATAXIA (Nervous system disorders) | 3 (3)
BALANCE DISORDER (Nervous system disorders) | 6 (6)
DIZZINESS (Nervous system disorders) | 12 (15)
HEADACHE (Nervous system disorders) | 17 (35)
HYPOAESTHESIA (Nervous system disorders) | 3 (3)
SEIZURE (Nervous system disorders) | 9 (11)
SOMNOLENCE (Nervous system disorders) | 20 (30)
ANXIETY (Psychiatric disorders) | 8 (8)
INSOMNIA (Psychiatric disorders) | 4 (4)
IRRITABILITY (Psychiatric disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
This trial was closed early after CVL-865-SZ-001 (NCT04244175) did not meet its primary objective

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04686786/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT04686786/SAP_001.pdf